CLINICAL TRIAL: NCT06587334
Title: the Clinical Effect of Nd: YAG Laser Assisted Periodontal Initial Therapy in Patients With Moderate to Severe Periodontitis: a Split-mouth, Randomized, Controlled Clinical Trial
Brief Title: the Clinical Effect of Nd: YAG Laser Assisted Periodontal Initial Therapy in Patients With Moderate to Severe Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1104
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis
Keywords: Nd: YAG Laser; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: The study adopts a split-mouth design with each subject serving as their own control. A random number method is used to determine whether the left or right half of the mouth will be assigned to the laser group, with the remaining half assigned to the control group. The laser group will receive SRP combined with Nd laser-assisted therapy, while the control group will receive SRP alone.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will receive SRP alone
  Interventions: Procedure: SRP
- Laser Group (Experimental): The laser group will receive SRP combined with Nd laser-assisted therapy
  Interventions: Procedure: Nd: YAG Laser Assisted SRP

INTERVENTIONS:
Procedure: SRP — SRP alone
  Arms: Control Group
Procedure: Nd: YAG Laser Assisted SRP — the patients receive SRP combined with Nd: YAG laser
  Arms: Laser Group

SUMMARY:
The goal of this clinical trial is to learn if Neodymium-Doped Yttrium Aluminum Garnet（Nd: YAG） Laser-assisted non-surgical periodontal treatment is effective in treating stage II/III periodontitis. It will also evaluate the safety and impact of the laser treatment. The main questions it aims to answer are:

1. Does Nd: YAG Laser treatment reduce probing depth, gingival inflammation, and clinical attachment loss more effectively than standard Scaling and root planing(SRP) therapy alone?
2. What changes in inflammatory markers and oxidative stress levels occur when patients receive laser-assisted therapy? Researchers will compare Nd: YAG Laser treatment to standard periodontal therapy alone to determine the effectiveness of the laser treatment.

Participants will:

1. Receive Nd: YAG Laser assisted therapy on one side of their mouth and standard therapy on the other side.
2. Visit the clinic at baseline, 6 weeks, and 3 months for follow-up assessments and tests.
3. Provide samples and have measurements taken of periodontal health and biomarkers of inflammation and oxidative stress.

DETAILED DESCRIPTION:
To investigate the clinical effect of Nd: YAG laser assisted non-surgical periodontal treatment on the patients with stage II / III periodontitis. This study included patients with stage II/III periodontitis who visited the Second Affiliated Hospital of Zhejiang University School of Medicine. Using a split-mouth design, the random number method was used to determine whether the left or right half of the subjects were in the laser group, and the remaining half were in the control group. All subjects underwent periodontal initial therapy, and the laser group received extra periodontal irradiation treatment using Nd: YAG laser. Before treatment, 6 weeks after treatment, and 3 months after treatment, the probing depth (PD), gingival index (GI), and clinical attachment loss (CAL) of all subjects were recorded. At the same time, the gingival crevicular fluid samples of thesubjects were collected using absorbent paper tips. The levels of Interleukin-6 (IL-6), Tumor necrosis factor-alpha (TNF-α), and Malondialdehyde (MDA) were measured using assay kits. Analyze and compare the changes in data before and after each group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years, with no gender restrictions.
* Diagnosed with stage II or III periodontitis according to the 2018 Classification of Periodontal and Peri-Implant Diseases and Conditions.
* In each of the four quadrants of the oral cavity, at least one tooth must have at least one site with a probing depth ≥5 mm, clinical attachment loss ≥2 mm, and bleeding on probing.
* Participants must provide informed consent and sign the informed consent form.

Exclusion Criteria:

* Fewer than 20 remaining teeth (10 pairs of opposing teeth) or a significant discrepancy in the number of remaining teeth between the left and right sides of the mouth.
* Patients who have undergone periodontal treatment within the past six months or are currently undergoing orthodontic treatment, which may affect periodontal health.
* Patients with systemic diseases that could influence the outcomes of periodontal treatment.
* Patients with severe infections, malignancies, or other major diseases affecting overall health.
* Pregnant or breastfeeding women.
* Individuals with a history of smoking.
* Patients who are unable to comply with or complete periodontal treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Probing depth，PD | Baseline，6 weeks，3months
  Probing depth refers to the distance from the gingival margin to the base of the periodontal pocket. It is measured using a periodontal probe at multiple sites around each tooth. A reduction in probing depth is indicative of periodontal health improvement following treatment.

SECONDARY OUTCOMES:
Gingival index，GI | Baseline，6 weeks，3months
  The Gingival Index is a clinical measure used to assess the severity of gingivitis based on the presence of inflammation, bleeding on probing, and changes in gingival color. It is scored on a scale from 0 (healthy gingiva) to 3 (severe inflammation). Lower scores post-treatment suggest improved gingival health.
Clinical attachment loss，CAL | Baseline，6 weeks，3months
  Clinical attachment loss is the measurement of the distance from the cemento-enamel junction (CEJ) to the base of the periodontal pocket. It reflects the extent of periodontal tissue destruction. A decrease in CAL indicates successful periodontal treatment and improved attachment of the tooth to the surrounding bone and tissue.
Concentration of interleukin-6（IL-6） | Baseline，6 weeks，3months
  Interleukin-6 is a pro-inflammatory cytokine measured in gingival crevicular fluid. It is used as a biomarker to assess the inflammatory response in periodontal tissues. Higher levels are associated with active inflammation, and a reduction post-treatment may indicate a successful anti-inflammatory effect of the therapy.
Concentration of tumor necrosis factor-alpha（TNF-α） | Baseline，6 weeks，3months
  Tumor necrosis factor-alpha is another key pro-inflammatory cytokine involved in the pathogenesis of periodontal disease. It is typically measured in gingival crevicular fluid. Similar to IL-6, elevated levels suggest active inflammation, while decreased levels post-treatment indicate a reduction in inflammatory activity.
Concentration of malondialdehyde（MDA） | Baseline，6 weeks，3months
  Malondialdehyde is a biomarker of oxidative stress, typically measured in gingival crevicular fluid. It reflects the extent of lipid peroxidation and cellular damage. Lower MDA levels after treatment suggest reduced oxidative stress and potential improvement in periodontal tissue health.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Tan, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Bian Z, Zhang H, Chen Y, Yang Y, Lin Q, Chen X, Chen L, Sun W, Tan J. Clinical effect of Nd:YAG laser-assisted non-surgical periodontal treatment on stage II/III periodontitis. J Dent. 2025 Nov;162:106056. doi: 10.1016/j.jdent.2025.106056. Epub 2025 Aug 26. PMID 40876623